CLINICAL TRIAL: NCT01169727
Title: Observational Study to Evaluate Health Status of Chronic Obstructive Pulmonary Disease (COPD) Patients in Response to Real-life Treatments in Thailand
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RTH-DUM-2009/2
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD and CCQ score; Changes in PEF,overall CCQ score
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate health status of uncontrolled Chronic Obstructive Pulmonary Disease (COPD) patients in response to treatments in clinical practice.

DETAILED DESCRIPTION:
MC MD

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male or non-pregnant female aged >40 years
3. A clinical diagnosis of COPD with FEV1/ FVC <0.70 and require combination or modified therapy
4. Smoke > 10 Pack Year

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Participation in a clinical study (precluding non-interventional study or registry) during the last 3 months

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care and Specialty care in 20 centers nationwide in Thailand
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in PEF and overall CCQ score | between the first visit and after 12 (plus or minus 1) weeks

SECONDARY OUTCOMES:
Difference of the changes of PEF and overall CCQ score comparing between various treatments | between the first visit and after 12 (plus or minus 1) weeks

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. Watchara Boonsawat, Principal Investigator — Khon Kaen University
Locations (20):
- Thailand (20):
  - Research Site, SaiMai, Bangkok
  - Research Site, Watana, Bangkok
  - Research Site, Maung, Changwat Chanthaburi
  - Research Site, Maung, Changwat Chiang Rai
  - Research Site, Muang, Changwat Chon Buri
  - Research Site, Muang, Changwat Khon Kaen
  - Research Site, Ongkharak, Changwat Nakhon Nayok
  - Research Site, Maung, Changwat Nonthaburi
  - Research Site, Muang, Changwat Phitsanulok
  - Research Site, Maung, Changwat Rayong
  - Research Site, Hat Yai, Changwat Songkhla
  - Research Site, Song Phi Nong, Changwat Suphan Buri
  - Research Site, Maung, Changwat Trang
  - Research Site, Maung, Chiang Mai
  - Research Site, Maung, Nakhon Sri Thammarat
  - Research Site, Maung, Nakhonratchasima
  - Research Site, Maung, Nakhonsawan
  - Research Site, Maung, Phuket
  - Research Site, Maung, Sakolnakorn
  - Research Site, Prannok, Bangkok